CLINICAL TRIAL: NCT03648086
Title: Efficacy, Safety of Intestinal Microbiota Transplantation for Nonalcoholic Fatty Liver Disease
Brief Title: Intestinal Microbiota Transplantation for Nonalcoholic Fatty Liver Disease
Acronym: NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017005
Record Dates: First submitted 2017-10-25; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2017-10

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: an open label, parallel study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT (Experimental): 30 non-alcoholic fatty liver disease（NAFLD） patients will be recruited for the study, which involved a 6 times intestinal microbiota transplant(IMT) and the time interval is generally 2 weeks.
  Interventions: Other: intestinal microbiota transplantation
- control (No Intervention): 30 non-alcoholic fatty liver disease(NAFLD) patients without any treatment

INTERVENTIONS:
Other: intestinal microbiota transplantation — Participants in Exprerimental group take 6 times IMT with 2-week intervals
  Other Names: IMT
  Arms: IMT

SUMMARY:
In China, with the improvement of living standards, there is a significant increase in the rate of prevalence of type 2 diabetes and hyperlipidemia, associated with Non-alcoholic fatty liver disease（NAFLD） which has gradually become a major public health problem in our country. The latest study found that intestinal microflora imbalance is closely correlated with NAFLD. In this subject, the investigators aim to explore whether intestinal microbiota transplantation(IMT) could reverse the change of intestinal microflora imbalance and has direct effects of NAFLD.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a significant health problem. With the trend of obesity and associated metabolic syndrome globally, nonalcoholic fatty liver disease has become a high incidence of liver disease in developed countries, the prevalence rate of NAFLD adult is about 10% ~ 30%. Therefore, effective prevention and treatment of NAFLD has important significance in improving people's quality of life and disease prognosis. The latest study found that intestinal microflora imbalance is closely correlated with NAFLD. When the structure of intestinal flora is destroyed, host energy absorption and storage of fat balance will be broken, with higher absorption of efficiency. At the same time, metabolic disorder expands. In this projects the investigators aim to re-establish a gut balance of intestinal microbiota through Standardized Intestinal Microbiota Transplantation for NAFLD. The CT ratio of liver/spleen, Fibroscan E value, general indicators, biochemical indicators will be used to assess the efficiency, durability and safety of Standardized IMT at the start and end of the projects.

ELIGIBILITY:
Inclusion Criteria:

* subjects with NAFLD(nonalcoholic fatty liver disease)
* aged 18-65
* 24≤BMI
* liver/spleen (L/S) ratio no more than 0.7 by CT scan

Exclusion Criteria:

* Alcoholic liver disease (ALD), chronic hepatitis C, autoimmune liver disease, Wilson's disease
* Drug treatment (tamoxifen, amiodarone, sodium valproate, methotrexate, glucocorticoids, etc.), total parenteral nutrition, inflammatory bowel disease, hypothyroidism, Cushing's syndrome, beta lipoprotein deficiency, IR related syndromes (lipid wasting diabetes mellitus, Mauriac syndrome), gastrointestinal surgery
* Hepatocellular carcinoma (HCC), biliary tract diseases and taking or taking chinese and western medicines that can lead liver enzymes elevation in the near future.
* Moderate and severe renal injuty(serum creatinine>2mg/dL or 177mmol/L), moderate and severe chronic obstructive pulmonary disease, severe hypertension, cerebrovascular accident, congestive heart failure, unstable angina pectoris.
* Antibiotics treatment in 7 days before recruited and unwilling to stop it, long-term lipid-lowering drugs, antidiabetic drugs and other liver protecting drugs treatment
* Antibiotics, other probiotics, gastrointestinal motility drugs and other preparation that may influence intestinal microbiota treatment
* Other serious diseases that may interfere the recruitment or affect the survival, such as cancer or acquired immune deficiency syndrome
* Mentally or legally disabled person
* Preparing for pregnancy
* Medical or social condition which in the opinion of the principal investigator would interfere with or prevent regular follow up
* Participating in other clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-14 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
The change of CT ratio of liver/spleen | 3 months, 6months
  CT imaging has been used to assess hepatic steatosis and has been validated in relation to liver biopsy .The ratio of liver to spleen (L/S ratio) for CT attenuation values is an index, with a L/S ratio<1 considered to represent fatty liver .The change of CT ratio of liver/spleen will be assessed at different time comparing with the baseline.

SECONDARY OUTCOMES:
biochemical indicators | 3 months, 6months
  Liver function such as ALT,AST,ALT/AST will be assessed at different time comparing with the baseline.
Fibroscan E value | 3 months, 6 months
  Fibroscan E value is a indicators for evaluating liver fibrosis.Changes will be assessed at different time comparing with the baseline.
Changes of gut microbiota | 3 months, 6months
  Alpha and Beta diversity of GI microbiota by High-throughput sequencing on baseline line and 3 months, 6months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Informed Consent Form (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT03648086/ICF_000.pdf
  • Study Protocol (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT03648086/Prot_001.pdf